CLINICAL TRIAL: NCT02681783
Title: PRedictive Factors and Changes From Treatment in Idiopathic Polypoidal Choroidal Vasuclopathy Versus Central Serous Chorioretinopathy Versus Neovascular Age Related Macular Degeneration With afLibercept
Brief Title: PRedictive Factors and Changes From Treatment in iPCV Versus CSR Versus nAMD With afLibercept
Acronym: PRaCTICAL
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Radha Kohly, Assistant Professor, University of Toronto, Sunnybrook Health Sciences Centre
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRaCTICAL 100-17
Record Dates: First submitted 2015-02-12; First posted 2016-02-12 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Central Serous Chorioretinopathy; Age Related Macular Degeneration; Idiopathic Poplypoidal Choroidal Vasculopathy
Keywords: aflibercept
MeSH Terms: conditions — Central Serous Chorioretinopathy; Macular Degeneration | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- neovascular AMD group with PED (Active Comparator): Patients in this group will be administered aflibercept intravitreal injection 2 mg (0.05 mL), administered at baseline, month 1, and month 2, for a total of 3 injections. Study will end for these patients at month 4, where no injection will be given. A clinical exam and OCT imaging will be performed each visit.
  Interventions: Drug: aflibercept
- CSR group with PED (Experimental): Patients in this group will be administered aflibercept intravitreal injection 2 mg (0.05 mL), administered at baseline, month 1, and month 2, for a total of 3 injections. Study will end for these patients at month 4, where no injection will be given. A clinical exam and OCT imaging will be performed each visit.
  Interventions: Drug: aflibercept
- iPCV group with PED (Experimental): Patients in this group will be administered aflibercept intravitreal injection 2 mg (0.05 mL), administered at baseline, month 1, and month 2, for a total of 3 injections. Study will end for these patients at month 4, where no injection will be given. A clinical exam and OCT imaging will be performed each visit.
  Interventions: Drug: aflibercept
- cataract patients (No Intervention): Patients diagnosed with cataracts requiring cataract surgery will serve as study controls. No intervention will be applied to these patients.

INTERVENTIONS:
Drug: aflibercept — Therapeutic/Pharmacological Classification: VEGF - Anti-neovascularization agent Route(s) of Administration: Intravitreal Injection Dosage Form: Solution 40 mg/ml Proposed Indication: Treatment of Pigment Epithelial Detachments (PEDs) associated with neovascular Age-related Macular Degeneration (nAMD), Central serous chorioretinopathy (CSR), and idiopathic Poplypoidal Choroidal Vasculopathy (iPCV).
  Other Names: Eylea
  Arms: CSR group with PED; iPCV group with PED; neovascular AMD group with PED

SUMMARY:
The presence of PEDs in nAMD, CSR and iPCV can present a diagnostic challenge in the elderly population; despite detailed diagnostic testing to differentiate these three conditions, misdiagnosis and mistreatment still occurs. One potential way of differentiating these three conditions might be to compare cytokine profiles in nAMD versus CSR versus iPCV. This information may be useful in creating a diagnostic aqueous cytokine and hormone profile to differentiate between nAMD, CSR and iPCV.

The primary goal of this study is to compare baseline aqueous cytokine and cortisol levels between nAMD, CSR, and iPCV patients and age-matched cataract controls. The secondary objective is to assess intra-group changes in visual and anatomical outcomes in nAMD, CSR and iPCV patients with PED treated with aflibercept and correlate these changes to baseline cytokines.

DETAILED DESCRIPTION:
The presence of Pigment Epithelial Detachments (PEDs) in neovascular Age-related Macular Degeneration (nAMD), Central serous chorioretinopathy (CSR) and idiopathic Poplypoidal Choroidal Vasculopathy (iPCV) can present a diagnostic challenge in the elderly population; despite detailed diagnostic testing to differentiate these three conditions, misdiagnosis and mistreatment still occurs. One potential way of differentiating these three conditions might be to compare cytokine profiles in nAMD versus CSR versus iPCV. In nAMD, growth factors and cytokines, such as vascular endothelial growth factor (VEGF), pigment epithelium derived factor (PEDF), interleukin 6 (IL-6) and placenta growth factor (PLGF) are known to play an important role in the development of CNV angiogenesis. Aqueous samples from CSR eyes have been analyzed for various growth factors and cytokines, where levels of interlukin (IL)-6, IL-8 and monocyte chemoattractant protein-1 do not differ from healthy controls, and platelet-derived growth factor (PDGF) levels appear to be lower than controls. In addition, there is evidence to demonstrate that CSR is associated with elevated cortisol serum levels. Cortisol has been analyzed in the aqueous humor of glaucoma and cataract patients; however, the presence of cortisol in aqueous humor in CSR patients has not yet been identified. One study comparing iPCV versus controls found elevated levels of IL-23. Cytokines have also been compared between nAMD and iPCV showing elevated levels of CRP and IL-10 in eyes with iPCV or nAMD. However, there have not been any studies yet comparing aqueous cytokine levels, including PLGF between iPCV, CSR, and nAMD patients. This information may be useful in creating a diagnostic aqueous cytokine and hormone profile to differentiate between nAMD, CSR and iPCV.

If left untreated, PEDs associated with nAMD, CSR, and iPCV may lead to the loss of central vision. We propose to compare the effectiveness of aflibercept in the treatment of PEDs associated with nAMD, CSR and iPCV.

The primary goal of this study is to compare baseline aqueous cytokine and cortisol levels between nAMD, CSR, and iPCV participants and age-matched cataract controls. We will not be looking at changes in cytokine levels after treatment. The secondary objective is to assess intra-group changes in visual and anatomical outcomes in nAMD, CSR and iPCV participants with PED treated with aflibercept and correlate these changes to baseline cytokines.

ELIGIBILITY:
Inclusion criteria for all study eye groups:

1. 18 years of age or older
2. Ability to provide signed informed consent
3. Capable of complying with study protocol and required diagnostic tests
4. Meets study eye criteria for each respective group (see Section 5 above)
5. Participants in the nAMD, CSR, and iPCV groups must use an acceptable method of birth control during this study and for 6 months following completion of the study. The participants in the control group will not be receiving IP and are not required to meet this inclusion criterion.

Exclusion criteria for all study eye groups:

1. Previous intraocular injections including anti-VEGF therapy or steroid medication, or macular laser for all groups
2. Any co-existing maculopathy or retinopathy in the study eye
3. Participants with a history of either type I or type II diabetes
4. Intraocular surgery in the study eye within the past 4 months
5. Currently on systemic steroid therapy in any form (drops, skin creams, inhalation/intranasal sprays, intravenous) or immunosuppression for the last 3 months
6. Participants on renal dialysis
7. Pregnant and nursing mothers
8. Participants who are hypersensitive to this drug, to any ingredient in the formulation, or to any component of the container.
9. Ocular or periocular infection
10. Active intraocular inflammation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Baseline aqueous humour cytokine levels in nAMD, CSR, and iPCV patients | 4 months from baseline intervention
  The primary outcome is to compare the baseline aqueous inflammatory cytokine levels (pg/ml) and baseline aqueous cortisol levels (pg/ml) through analyzing anterior chamber aqueous fluid in patients with nAMD, CSR, and iPCV patients receiving aflibercept intravitreal injections, and compare with the aquueous fluid of age-matched control patients undergoing cataract surgery.

SECONDARY OUTCOMES:
Assessment of the intra-group changes in best-corrected visual acuity using Snellen eye charts after aflibercept treatment in patients with nAMD, CSR, and iPCV for 4 months | 4 months from baseline intervention
  To assess the intra-group changes in best-corrected visual acuity using Snellen eye charts after aflibercept treatment in patients with nAMD, CSR, and iPCV for 4 months
Assessment of the intra-group changes in anatomical changes via OCT imaging from baseline after aflibercept treatment in patients with nAMD, CSR, and iPCV for 4 months | 4 months from baseline intervention
  To assess the intra-group changes in anatomical changes via OCT imaging from baseline after aflibercept treatment in patients with nAMD, CSR, and iPCV for 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Radha P. Kohly, MD PhD FRCSC, Principal Investigator — Sunnybrook Health Sciences Center
Locations (1):
- Sunnybrook Research Institute, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided